CLINICAL TRIAL: NCT04856904
Title: Evaluation of the Risk of Atrophic Acne Scar Formation During Treatment of Acne Vulgaris Subjects With Trifarotene 50 μg/g Cream Versus Vehicle Cream Over 24 Weeks
Brief Title: Study of Trifarotene Cream to Assess Risk of a Trophic Acne Scar Formation
Acronym: START
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.202395; 2020-006050-51 (EudraCT Number)
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2023-12

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Trifarotene; AKLIEF®; CD5789
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trifarotene Vehicle Cream (Placebo Comparator)
  Interventions: Drug: Trifarotene Vehicle Cream
- Trifarotene (CD5789) 50 mcg/g Cream (Experimental)
  Interventions: Drug: Trifarotene Cream

INTERVENTIONS:
Drug: Trifarotene Cream — Participants will apply a thin a layer of trifarotene (CD5789) 50 mcg/g cream to the face once daily, in the evening for 24 weeks
  Other Names: AKLIEF®
  Arms: Trifarotene (CD5789) 50 mcg/g Cream
Drug: Trifarotene Vehicle Cream — Participants will apply a thin a layer of trifarotene vehicle cream to the face once daily, in the evening for 24 weeks
  Arms: Trifarotene Vehicle Cream

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of trifarotene 50 microgram per gram (mcg/g) cream compared to its vehicle on the risk of formation of atrophic acne scars after 24 weeks of treatment in facial acne participants assessed by atrophic acne scars count.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant with clinical diagnosis of acne vulgaris on the face as defined by (excluding the nose and middle zone of approximately 2 centimeter [cm]):

  1. Investigator's Global Assessment (IGA) score of 3 (Moderate) or 4 (Severe), with the same score on both sides of the face; and
  2. A minimum of 20 inflammatory lesions (papules and pustules) in total with at least 10 on each side; and
  3. No more than 2 nodules (greater than or equal to [>=] 1 cm in diameter) on the face; and
  4. A minimum of 10 atrophic acne scars in total (>2 mm)
* Participant with a symmetrical number of the following lesions/scars on the whole face:

  1. Inflammatory and non-inflammatory lesions; and
  2. Atrophic acne scars (minimum of 4 scars per half-face)
* The participant is a female of non-childbearing potential
* If a female of childbearing, potential uses oral contraceptives that are also approve for treating acne vulgaris
* Other protocol defined inclusion criteria could apply

Key Exclusion Criteria:

* Participant with acne conglobata, acne fulminans, secondary acne, nodulocystic acne and acne requiring systemic treatment
* Participant with any acne cyst on the face or with more than 3 excoriated acne lesions
* Participant with known active or chronic allergies or suspected allergy to trifarotene or excipients of the formulation
* Participant with facial dermal conditions (for example, tattoo, skin abrasion, eczema, sunburned skin, scars, nevi, etc.) that may interfere with study assessments in the opinion of the investigator
* Participant with known impaired hepatic or renal functions, based on medical history

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (15):
  - Galderma Investigational Site #8873, Scottsdale, Arizona
  - Galderma Investigational Site #8447, Fort Smith, Arkansas
  - Galderma Investigational Site #8608, Santa Monica, California
  - Galderma Investigational Site #9928, Boynton Beach, Florida
  - Galderma Investigational Site #8295, Miami, Florida
  - Galderma Investigational Site #8883, Miramar, Florida
  - Galderma Investigational Site #8189, Snellville, Georgia
  - Galderma Investigational Site #8367, Arlington Heights, Illinois
  - Galderma Investigational Site #8838, Darien, Illinois
  - Galderma Investigational Site #8601, Metairie, Louisiana
  - Galderma Investigational Site #9936, New Orleans, Louisiana
  - Galderma Investigational Site #8108, Las Vegas, Nevada
  - Galderma Investigational Site #8881, Stony Brook, New York
  - Galderma Investigational Site #8886, Sugarloaf, Pennsylvania
  - Galderma Investigational Site #9920, Arlington, Texas
- Canada (2):
  - Galderma Investigational Site #9918, Peterborough, Ontario
  - Galderma Investigational Site #9927, Saint-Jérôme, Quebec
- Galderma Investigational Site #6167, Nantes, France

REFERENCES:
- [Derived] Schleicher S, Moore A, Rafal E, Gagne-Henley A, Johnson SM, Dhawan S, Chavda R, York JP, Sforzolini B, Holcomb K, Ablon G, Del Rosso J, Dreno B. Trifarotene Reduces Risk for Atrophic Acne Scars: Results from A Phase 4 Controlled Study. Dermatol Ther (Heidelb). 2023 Dec;13(12):3085-3096. doi: 10.1007/s13555-023-01042-7. Epub 2023 Oct 15. PMID 37838987

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 sites in the United States, Canada, and France.
Pre-assignment Details: A total 121 participants were enrolled in this study. All participants were randomized (left face versus right face) to apply trifarotene cream and trifarotene vehicle cream for an intra-individual, split-face comparison.
Units Other Than Participants: half faces
Groups:
- Trifarotene 50mcg/g Cream: Participants applied a thin layer of trifarotene cream to half of their face topically once daily for up to 24 weeks.
- Trifarotene Vehicle Cream: Participants applied a thin layer of trifarotene vehicle cream to another half of their face topically once daily for up to 24 weeks.
Period: Overall Study
Arm/Group | Trifarotene 50mcg/g Cream | Trifarotene Vehicle Cream
Started | 121; 121 half faces | 121; 121 half faces
Completed | 99; 99 half faces | 99; 99 half faces
Not Completed | 22; 22 half faces | 22; 22 half faces
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 13 | 13
Not completed — Adverse Event | 1 | 1
Not completed — Non-compliance with study drug | 1 | 1
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized partcipants.
Groups:
- All Acne Vulgaris Participants: All participants applied a thin layer of trifarotene 50 mcg/g cream to half of their face and trifarotene vehicle cream to another half of their face topically once daily for up to 24 weeks.
Arm/Group | All Acne Vulgaris Participants
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (5.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 95
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 97
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: count of participants]
  Canada | 9
  United States | 110
  France | 2
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Skin Type I = White; very fair, red or blonde hair blue eyes; freckles; Always burns, never tans Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes; Usually burns, tans with difficulty Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily Skin Type VI = Black; Never burns, tans very easily
  Participants
    Type I | 7
    Type II | 43
    Type III | 31
    Type IV | 26
    Type V | 11
    Type VI | 3

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Total Atrophic Acne Scar Count Per Half Face at Week 24
Description: The scars were counted according to their size defined in two categories using 2 millimeter (mm) and 4 mm punch biopsy tools for size classification: 1) atrophic scars 2 to 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types; 2) atrophic scars greater than (>) 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types. Each type of atrophic acne scar was counted separately for each half-face by the evaluator for following regions: right forehead, right cheek, right side of the chin, left forehead, left cheek and left side of the chin. To obtain the total number of atrophic scars per half-face, atrophic acne scar counts for each half-face was added.
Time Frame: Baseline, Week 24
Population: ITT population included all randomized participants.
Measure: Mean (Standard Error); unit: atrophic acne scars
Arm/Group | Trifarotene 50mcg/g Cream | Trifarotene Vehicle Cream
Number analyzed (Participants) | 121 | 121
atrophic acne scars | -5.9 (0.51) | -2.7 (0.37)
Statistical Analysis 1: Comparison: Trifarotene 50mcg/g Cream vs Trifarotene Vehicle Cream; Test type: Superiority; p < 0.0001, Student's t-test for paired samples; Bilateral difference = -3.2, 95% CI 2-sided [-4.4 to -2], Standard Error of Mean 0.6

2. Secondary Outcome: Absolute Change From Baseline in Total Atrophic Acne Scar Count Per Half-Face up to Week 20
Description: The scars were counted according to their size defined in two categories using 2 mm and 4 mm punch biopsy tools for size classification: 1) atrophic scars 2 to 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types; 2) atrophic scars > 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types. Each type of atrophic acne scar was counted separately for each half-face by the evaluator for following regions: right forehead, right cheek, right side of the chin, left forehead, left cheek and left side of the chin. To obtain the total number of atrophic scars per half-face, atrophic acne scar counts for each half-face was added.
Time Frame: Baseline, up to Week 20
Population: ITT population included all randomized participants.
Measure: Mean (Standard Error); unit: atrophic acne scars
Arm/Group | Trifarotene 50mcg/g Cream | Trifarotene Vehicle Cream
Number analyzed (Participants) | 121 | 121
atrophic acne scars
  Change at Week 1 | -0.3 (0.21) | -0.3 (0.16)
  Change at Week 2 | -0.9 (0.26) | -0.4 (0.11)
  Change at Week 4 | -1.5 (0.27) | -0.7 (0.18)
  Change at Week 8 | -2.5 (0.30) | -1.1 (0.30)
  Change at Week 12 | -3.8 (0.37) | -1.7 (0.32)
  Change at Week 16 | -4.4 (0.40) | -1.7 (0.47)
  Change at Week 20 | -5.0 (0.47) | -2.5 (0.33)
Statistical Analysis 1: Comparison: Trifarotene 50mcg/g Cream vs Trifarotene Vehicle Cream; Week 1: Trifarotene 50 mcg/g, vehicle cream; Test type: Superiority; p = 0.9476, Student's t-test for paired samples; Bilateral difference = 0, 95% CI 2-sided [-0.3 to 0.3], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Trifarotene 50mcg/g Cream vs Trifarotene Vehicle Cream; Week 2: Trifarotene 50 mcg/g, vehicle cream; Test type: Superiority; p = 0.0248, Student's t-test for paired samples; Bilateral difference = -0.6, 95% CI 2-sided [-1.1 to -0.1], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: Trifarotene 50mcg/g Cream vs Trifarotene Vehicle Cream; Week 4: Trifarotene 50 mcg/g, vehicle cream; Test type: Superiority; p = 0.0072, Student's t-test for paired samples; Bilateral difference = -0.8, 95% CI 2-sided [-1.4 to -0.2], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Trifarotene 50mcg/g Cream vs Trifarotene Vehicle Cream; Week 8: Trifarotene 50 mcg/g, vehicle cream; Test type: Superiority; p < 0.0001, Student's t-test for paired samples; Bilateral difference = -1.4, 95% CI 2-sided [-2.1 to -0.7], Standard Error of Mean 0.35
Statistical Analysis 5: Comparison: Trifarotene 50mcg/g Cream vs Trifarotene Vehicle Cream; Week 12: Trifarotene 50 mcg/g, vehicle cream; Test type: Superiority; p < 0.0001, Student's t-test for paired samples; Bilateral difference = -2.1, 95% CI 2-sided [-2.9 to -1.3], Standard Error of Mean 0.41
Statistical Analysis 6: Comparison: Trifarotene 50mcg/g Cream vs Trifarotene Vehicle Cream; Week 16: Trifarotene 50 mcg/g, vehicle cream; Test type: Superiority; p < 0.0001, Student's t-test for paired samples; Bilateral difference = -2.7, 95% CI 2-sided [-3.8 to -1.6], Standard Error of Mean 0.56
Statistical Analysis 7: Comparison: Trifarotene 50mcg/g Cream vs Trifarotene Vehicle Cream; Week 20: Trifarotene 50 mcg/g, vehicle cream; Test type: Superiority; p < 0.0001, Student's t-test for paired samples; Bilateral difference = -2.5, 95% CI 2-sided [-3.5 to -1.5], Standard Error of Mean 0.53

ADVERSE EVENTS:
Time Frame: From screening up to Week 28
Description: The safety (SAF) population included the ITT population participants who applied the study drug at least once.
Arm/Group | Trifarotene 50mcg/g Cream | Trifarotene Vehicle Cream | All Acne Vulgaris Participants
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/121 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/121 | 0/121
Other Adverse Events (participants affected / at risk) | 7/121 | 3/121 | 33/121
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trifarotene 50mcg/g Cream (N=121) | Trifarotene Vehicle Cream (N=121) | All Acne Vulgaris Participants (N=121)
COVID-19 (Infections and infestations) | 0 | 0 | 10
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Skin tightness (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 2
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Adverse reaction (General disorders) | 1 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Vaccination site pain (General disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT04856904/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT04856904/SAP_001.pdf